CLINICAL TRIAL: NCT01199185
Title: Targeted Approaches to Weight Control for Young Adults
Brief Title: Treating Adults at Risk for Weight Gain With Interactive Technology
Acronym: TARGIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01HL096628 (NIH)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Smoking; Body Weight
MeSH Terms: conditions — Smoking; Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tobacco Quitline Group (Active Comparator)
  Interventions: Behavioral: Smoking Cessation
- Tobacco Quitline plus Interactive Technology Group (Experimental)
  Interventions: Behavioral: Smoking Cessation plus Weight Loss

INTERVENTIONS:
Behavioral: Smoking Cessation — All participants will receive a smoking cessation intervention via the Proactive TARGIT Quit Line. Participants will receive access to the TARGIT Smoking Cessation Handbook which will be a useful tool to guide them through the quitting process and highlight the major points reviewed in all counseling sessions. As part of TARGIT all participants will receive nicotine replacement therapy (NRT).
  Arms: Tobacco Quitline Group
Behavioral: Smoking Cessation plus Weight Loss — All participants will receive a smoking cessation intervention via the Proactive TARGIT Quit Line. Participants will receive access to the TARGIT Smoking Cessation Handbook which will be a useful tool to guide them through the quitting process and highlight the major points reviewed in all counseling sessions. As part of TARGIT all participants will receive nicotine replacement therapy (NRT). Participants in the Intervention Group will also receive a Behavioral Weight Loss/ Weight Gain Prevention Intervention delivered via interactive technology. The Intervention group will receive 16 weekly webinar sessions beginning 7 weeks after randomization via Cisco WebEx. The webinar sessions will present the behavioral weight loss/ weight gain prevention program. After the 16 weekly sessions, the webinar sessions will then be scheduled monthly for the next 6 months then quarterly thereafter for 12 months.
  Arms: Tobacco Quitline plus Interactive Technology Group

SUMMARY:
Obesity represents a chronic disease associated with significant cardiovascular disease (CVD) morbidity and mortality. Weight gain in young adults adversely impacts the development of CVD risk factors. Further, there is a clear relationship between weight loss in obese persons and reduction in these CVD risk factors. Unfortunately, young adults are at high risk for weight gain. Although the scientific literature contains a number of reports regarding successful weight loss efficacy studies, young adults are typically underrepresented.

Cigarette smoking is the leading preventable cause of morbidity and mortality, but quitting smoking frequently results in significant weight gain. Proactive tobacco quit lines using behavioral smoking cessation interventions combined with nicotine replacement therapy (NRT) have been shown to help persons quit smoking. However, concerns about post-cessation weight gain have been reported as a significant barrier to quitting for many smokers particularly young adults.

If an efficacious behavioral weight loss program could be combined with an efficacious behavioral smoking cessation program that prevented or significantly attenuated post-cessation weight gain, then a large public health benefit may result. Such a combined weight loss/ weight gain prevention / smoking cessation program that used targeted intervention strategies to young adults, removed barriers to participation, and utilize interactive technology should be appealing to this age group. To date such a combined program has not been tested in young adult cigarette smokers. Therefore, the objective of this clinical trial is to develop and test a behavioral weight loss / weight gain prevention intervention delivered through interactive technology that can be used in conjunction with an efficacious tobacco quit line. A total of 330 participants will be necessary to adequately address the following specific aims.

ELIGIBILITY:
Inclusion Criteria:

The selection criteria for the clinical trial are designed to include a wide range of participants such that the study sample will be representative of the broader U.S. population of the Memphis metropolitan area. Those who might be at risk of adverse outcomes from the study interventions will be excluded (see exclusion criteria). All participants will give voluntary consent at the screening visit by signing an informed consent statement which has been approved by the Institutional Review Board (IRB). We will encourage the participation of women and minorities. The study will be open to all persons of any race or gender who are:

1. *18 to 35 years old
2. BMI > 22 kg / m2
3. Self report smoking > 10 cigarettes each day
4. Have access to a telephone and the internet
5. Demonstrate ability to access a specific web site
6. Demonstrate ability to receive and respond to email
7. Willing to accept random assignment
8. *Intending to be available for a 24 month intervention
9. *At risk for weight gain (e.g. plan to quit smoking)

Exclusion Criteria:

Persons will be excluded from the TARGIT study for the following:

1. *Current participation in a commercial weight loss program (e.g. Weight Watchers, Jenny Craig, etc.), current use of a prescription weight loss medication, planned weight loss surgery within the next 24 months (e.g. gastric bypass, lap band, or liposuction), current or planned enrollment in another diet / physical activity / weight loss study
2. Currently meet recommendations for physical activity (i.e., 30 minutes or more of moderate physical activity per day on the majority of days each week - 150 minutes or more each week)
3. *History of cerebral, coronary, or peripheral vascular disease, or serious uncontrolled cardiac arrhythmia, revascularization procedure or uncontrolled congestive heart failure in the past 6 months
4. Current substance abuse (includes alcohol use in excess of 21 drinks a week)
5. Uncontrolled hypertension as defined as BP > 140/90 mm Hg
6. Presence of an unstable psychiatric condition or use of anti-psychotic drugs
7. History of significant kidney disease or liver disease
8. History of uncontrolled thyroid disease or pheochromocytoma
9. Current use of a medication that may interfere with primary study endpoints (e.g. a weight loss medication such as Orlistat, etc) or that may increase the risk of side effects from the study intervention that can not be discontinued
10. Severe uncontrolled asthma, bronchitis, or emphysema that precludes exercise
11. Resting heart rate > 100
12. *Malignancy in the last 5 years (except non-melanoma skin cancer)
13. Plans to move from the Memphis metropolitan area in the next two years
14. Current participation in another clinical trial
15. *Other medical or behavioral factors, that in the judgment of the Principal Investigator, may interfere with study participation or the ability to follow the intervention protocol
16. *History of diabetes treated with a medication that may cause hypoglycemia such as insulin or an oral hypoglycemic agent
17. Known allergy or sensitivity to the nicotine patch
18. *Currently pregnant or gave birth within the last 6 months, currently lactating or breast feeding within the last 3 months, actively planning pregnancy within the next 24 months
19. *BMI < 18.5 kg / m2 or > 40 kg / m2
20. *Have a household member on study staff
21. *Current treatment for an eating disorder
22. *Unable to provide informed consent
23. *Regular use of a systemic steroids defined as taking the medication most days of the week
24. *Use of medications to treat attention deficit disorder (ADD) or attention deficit hyperactivity disorder (ADHD)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Estimated)
Dates: Start 2009-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 24 months after randomization

SECONDARY OUTCOMES:
Smoking status | 24 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Karen Johnson, MD, MPH, Principal Investigator — University of Tennessee
Locations (1):
- Department of Preventive Medicine, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Johnson KC, Thomas F, Richey P, Tran QT, Tylavsky F, Miro D, Coday M. The Primary Results of the Treating Adult Smokers at Risk for Weight Gain with Interactive Technology (TARGIT) Study. Obesity (Silver Spring). 2017 Oct;25(10):1691-1698. doi: 10.1002/oby.21968. PMID 28948720